CLINICAL TRIAL: NCT04664452
Title: Current Status of Utilization an Surgeons' View of Porcine Derived Medical Products: an International Survey
Brief Title: Current Status of Porcine Derived Products in Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Elvan Onur Kirimker, Attending Surgeon at Dept of Surgery, Ankara University
Other Study IDs: PORCINE2020
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Ethics, Narrative
Keywords: porcine; ethics; informed consent; biological graft
MeSH Terms: conditions — Narration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Participants will be asked to fill the questionnaire

SUMMARY:
Porcine derived products are being used as biological grafts in mainly in orthopedic surgery, neurosurgery, cardiovascular surgery and general surgery. It is well known that consuming pork or porcine products are prohibited in some religions or divisions of religions. It may be a tender point for patients undergoing surgery in which porcine derived products are utilized.In this survey study we aimed to determine the level of awareness and perception of surgeons with an international anquette. The study will also reveal the choices of surgeons about this issue both in elective and emergency procedures

DETAILED DESCRIPTION:
In the survey study an online anquette form will be sent through online surgery networks both professional and social media. The questionnaire will not include questions defining the responders individually. The questions are related to frequency of utilization of porcine derived products in surgery, surgeons' level of awareness about utilization of porcine products, surgeons' level of religiousity and surgeons' choices about porcine derived product utilization and consent of patients. After collection of responses the data will be analyzed to discover current status of porcine derived surgical product utilization and surgeons' perception about the issue. The anquette will be distributed worldwide to surgeons in different branches of surgery. Literature seems to be lacking of that kind of study

ELIGIBILITY:
Inclusion Criteria:

* Being volunteer and responder of at least 80% of the study questionnaire

Exclusion Criteria:

* Responding less than 80% of the questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Specialist of any branch of surgery excluding pathology and anesthesiology
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-05 (Estimated); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Surgeons' awareness of utilization of porcine derived products in surgery | 2 month
  Frequency of awareness and experience on porcine derived medical products
Surgeons' choice about utilization of porcine derived products in surgery | 2 month
  Choices of surgeons on specific scenarios in the questionnaire

SECONDARY OUTCOMES:
Relationship of porcine derived product utilization according to religious/phlosophical belief | 2 month
  Choices of surgeons according to Religiousness Scale of Altemayer
Surgeons' choice about informing patients about porcine derived products | 2 month
  What ar e the choices of surgeons about informing patients and their relatives in described scenarios in the questionnaire

IPD SHARING:
Plan to Share IPD: No
Only study protocol and results will be shared on the clinicaltrials.gov